CLINICAL TRIAL: NCT07053111
Title: The Counselor Led Resident Wellness Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23347451
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Burnout, Healthcare Workers; Anxiety; Wellness Program; Depression Not Otherwise Specified
Keywords: Randomized Controlled Trial; Resident Wellness; Counselor
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselor Wellness Intervention (Experimental): Evidenced based, counselor lead wellness intervention that will provide psychoeducational peer support/peer process groups. Topics may include: work/life balance, resilience building, stress management, self- care practices, imposter syndrome, psychological effects, compassion fatigue, peer support, and mindfulness practices. Other evidence based therapeutic concepts, such as Cognitive Behavior Therapy (CBT) and Dialectical Behavior Therapy (DBT), may also be introduced as appropriate. The intervention group will also receive standard access to all mental health and wellness interventions at the university.
  Interventions: Behavioral: Wellness Intervention
- Control Group (No Intervention): Standard access to all mental health and wellness interventions at the university.

INTERVENTIONS:
Behavioral: Wellness Intervention — Licensed counselors will provide evidence based curricula on the following: work/life balance, resilience building, stress management, self- care practices, imposter syndrome, psychological effects, compassion fatigue, peer support, and mindfulness practices.
  Arms: Counselor Wellness Intervention

SUMMARY:
Residency is a challenging time in a physician's career. The investigators hope this study will provide a new wellness support model for residency programs to use for resident physicians. The purpose of this study is to examine the impact of a wellness support model for residency programs that is lead by licensed counselors. The investigators expect that participating resident physicians will feel and perform better in their job and your life with this additional support.

DETAILED DESCRIPTION:
Residency training has been identified as a challenging time in a physician's career. Prior studies have identified the positive effects of wellness support services on resident and attending physician wellbeing and burnout. A recent systematic review in PLoS One identified only one study in which counselors or psychologists, as opposed to peer mentors or other professionals including coaches, were utilized for the mental health wellness intervention. These studies show a benefit for some but not all metrics studied. Professional therapists may have additional skills or insight that may enhance wellness interventions. To help improve physician wellness at the University Health (UNR Plumas) Clinic, the investigators have developed an evidence based counselor wellness support group. The study will be a parallel group randomized controlled trial that seeks to build upon the above literature but also introduce additional novel components. Specifically, the study will utilize trained mental health counselors, instead of online or in person coaches or trained peer support, to provide in person physician wellness services to resident physicians. It will track the efficacy of a longitudinal, evidence-based curriculum by collecting data on wellness, depression, and anxiety using standard metrics, with the goal of increasing physician wellness in a cost-effective manner.

ELIGIBILITY:
Inclusion Criteria:

-All internal medicine residents at the University of Nevada, Reno whose continuity clinic site is the University Health (UNR Plumas) Clinic for the 2025-2026 academic year will be offered the opportunity to participate.

Exclusion Criteria:

* Must be a UNR internal medicine resident as described above
* Residents must be interested/willing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The World Health Organization-Five Well-Being Index (WHO-5) | Approximately 10 months
  The WHO-5 is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being. Specifically, a score of 0 indicates the participant taking the survey has "At no time" experienced the statement in question, while a score of 5 indicates the participant experiences the statement "All of the time." A gradient of numbers in between 0-5 represents increasing in frequency of the given experience. The instrument has been translated into over 30 languages.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ - 9) | ~10 months
  Graded measurement of general depression severity. Participants answer 9 questions with scores from 0 (not at all) to 3 (nearly every day) for each question to determine depression severity. Higher numbers indicate higher possible depression severity.
GAD 7 | ~10 months
  Seven question general anxiety metric. Participants rate questions from 0 (not at all) to 3 (nearly every day) to give a general measure of anxiety severity. Higher numbers indicate higher anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kandel, DO, Principal Investigator — University of Nevada, Reno
Locations (1):
- University Health Internal Medicine Clinic, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Eskander J, Rajaguru PP, Greenberg PB. Evaluating Wellness Interventions for Resident Physicians: A Systematic Review. J Grad Med Educ. 2021 Feb;13(1):58-69. doi: 10.4300/JGME-D-20-00359.1. Epub 2020 Dec 31. PMID 33680302
- [Background] Underdahl L, Ditri M, Duthely LM. Physician Burnout: Evidence-Based Roadmaps to Prioritizing and Supporting Personal Wellbeing. J Healthc Leadersh. 2024 Jan 4;16:15-27. doi: 10.2147/JHL.S389245. eCollection 2024. PMID 38192639
- [Background] Boet S, Etherington C, Dion PM, Desjardins C, Kaur M, Ly V, Denis-LeBlanc M, Andreas C, Sriharan A. Impact of coaching on physician wellness: A systematic review. PLoS One. 2023 Feb 7;18(2):e0281406. doi: 10.1371/journal.pone.0281406. eCollection 2023. PMID 36749760
- [Background] Mann A, Shah AN, Thibodeau PS, Dyrbye L, Syed A, Woodward MA, Thurmon K, Jones CD, Dunbar KS, Fainstad T. Online Well-Being Group Coaching Program for Women Physician Trainees: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2335541. doi: 10.1001/jamanetworkopen.2023.35541. PMID 37792378
- [Background] Palamara K, Chu JT, Chang Y, Yu L, Cosco D, Higgins S, Tulsky A, Mourad R, Singh S, Steinhauser K, Donelan K. Who Benefits Most? A Multisite Study of Coaching and Resident Well-being. J Gen Intern Med. 2022 Feb;37(3):539-547. doi: 10.1007/s11606-021-06903-5. Epub 2021 Jun 7. PMID 34100238
- [Background] Solms L, van Vianen A, Koen J, Theeboom T, de Pagter APJ, De Hoog M; Challenge & Support Research Network. Turning the tide: a quasi-experimental study on a coaching intervention to reduce burn-out symptoms and foster personal resources among medical residents and specialists in the Netherlands. BMJ Open. 2021 Jan 25;11(1):e041708. doi: 10.1136/bmjopen-2020-041708. PMID 33495254
- [Background] Sofka S, Lerfald N, Reece J, Davisson L, Howsare J, Thompson J. Universal Well-Being Assessment Associated With Increased Resident Utilization of Mental Health Resources and Decrease in Professionalism Breaches. J Grad Med Educ. 2021 Feb;13(1):83-88. doi: 10.4300/JGME-D-20-00352.1. Epub 2020 Dec 31. PMID 33680305
- [Background] Raimo J, LaVine S, Spielmann K, Akerman M, Friedman KA, Katona K, Chaudhry S. The Correlation of Stress in Residency With Future Stress and Burnout: A 10-Year Prospective Cohort Study. J Grad Med Educ. 2018 Oct;10(5):524-531. doi: 10.4300/JGME-D-18-00273.1. PMID 30386477
- [Background] Salyers MP, Bonfils KA, Luther L, Firmin RL, White DA, Adams EL, Rollins AL. The Relationship Between Professional Burnout and Quality and Safety in Healthcare: A Meta-Analysis. J Gen Intern Med. 2017 Apr;32(4):475-482. doi: 10.1007/s11606-016-3886-9. Epub 2016 Oct 26. PMID 27785668
- [Background] Neumann M, Edelhauser F, Tauschel D, Fischer MR, Wirtz M, Woopen C, Haramati A, Scheffer C. Empathy decline and its reasons: a systematic review of studies with medical students and residents. Acad Med. 2011 Aug;86(8):996-1009. doi: 10.1097/ACM.0b013e318221e615. PMID 21670661
- [Background] Harvey SB, Epstein RM, Glozier N, Petrie K, Strudwick J, Gayed A, Dean K, Henderson M. Mental illness and suicide among physicians. Lancet. 2021 Sep 4;398(10303):920-930. doi: 10.1016/S0140-6736(21)01596-8. PMID 34481571